CLINICAL TRIAL: NCT03766646
Title: Preoxygenation With High Flow Nasal Oxygenation Using Optiflow - Does Speech Have an Effect on The End Tidal Oxygen Achieved When Compared to Closed Mouth Nasal Breathing?
Brief Title: Preoxygenation With Optiflow™ - the Effect of Speech on Lung Oxygenation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RHM CR10369
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Results first posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Unrecognized Condition
Keywords: Optiflow; High Flow Nasal Oxygen; Preoxygenation; Speech
MeSH Terms: conditions — Speech

STUDY DESIGN:
Intervention Model Description: Patients were assigned to either the 'Speech' arm or 'Non-speech' arm of the study
Masking Description: After recruitment, patients were randomised into one of two arms, speech or non-speech. Both the investigator and the participant were aware of the intervention assigned
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Speech (Experimental): Participants were asked to read a standardised script aloud for 3 minutes whilst receiving oxygen from the Optiflow device. At the end of 3 minutes End Tidal Oxygen was measured and recorded.
  Interventions: Device: Optiflow
- Non-speech (Active Comparator): Participants were asked to breathe in and out of their nose for 3 minutes, with a closed mouth, whilst receiving oxygen from the Optiflow device. At the end of 3 minutes End Tidal Oxygen was measured and recorded.
  Interventions: Device: Optiflow

INTERVENTIONS:
Device: Optiflow — 45l.min oxygen
  Other Names: HFNO, High Flow Nasal Oxygen

SUMMARY:
If a patient speaks during the process of preoxygenation with high-flow nasal oxygen via the Optiflow™ system, is the efficacy reduced as measured by end-tidal lung oxygen content?

DETAILED DESCRIPTION:
This is a randomised controlled trial on 34 patients undergoing routine elective surgery at the Princess Anne Hospital, Southampton. The study will take place from September 2018 to January 2019 and involve preoxygenating all participants for three minutes using the Optiflow™ device. During this time, participants will be instructed to either read aloud a standardised text or to breathe through their nose with a closed mouth. At the end of 3 minutes, the primary outcome, ETO2, will be measured and recorded.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-35, ASA category 1 or 2

Exclusion Criteria:

* Inability to read/ follow instructions, Heavily sedated

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2018-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Butler, Principal Investigator — Unvistery Hospital Southampton
Locations (1):
- University Hospital Southampton, Southampton, Hants, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Speech | Non-speech
Started | 19 | 15
Completed | 18 | 12
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Speech | Non-speech | Total
Number analyzed (Participants) | 19 | 15 | 34
Age, Categorical [Count of Participants; unit: Participants] — Population: Participants not suitable for analysis
  Participants
    number analyzed (Participants) | 18 | 12 | 30
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 18 | 12 | 30
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Participant withdrawal/ unsuitable for analysis
  Participants
    number analyzed (Participants) | 18 | 12 | 30
    Female | 18 | 12 | 30
    Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Median (Full Range); unit: kg.m-2] | 27.0 [20.3 to 31.8] | 26.5 [21.1 to 35.4] | 26.7 [20.3 to 35.4]

OUTCOME MEASURES:

1. Primary Outcome: End Tidal Oxygen Fraction
Description: Oxygen fraction in first expired breath post preoxygenation
Time Frame: At the end of 3 minutes preoxygenation
Measure: Mean (Standard Deviation); unit: percentage of End-Tidal Oxygen Fraction
Arm/Group | Speech | Non-speech
Number analyzed (Participants) | 18 | 12
percentage of End-Tidal Oxygen Fraction | 43.9 (15.4) | 81.9 (8.3)

ADVERSE EVENTS:
Groups:
- Speech: Participants were asked to read a standardised script aloud for 3 minutes whilst receiving oxygen from the Optiflow device. At the end of 3 minutes End Tidal Oxygen was measured and recorded.
  Optiflow: 45l.min oxygen
  All-Cause Mortality, Serious Adverse Events, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
- Non-speech: Participants were asked to breathe in and out of their nose for 3 minutes, with a closed mouth, whilst receiving oxygen from the Optiflow device. At the end of 3 minutes End Tidal Oxygen was measured and recorded.
  Optiflow: 45l.min oxygen
  All-Cause Mortality, Serious Adverse Events, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Speech | Non-speech
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/46/NCT03766646/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-17): https://cdn.clinicaltrials.gov/large-docs/46/NCT03766646/SAP_001.pdf